CLINICAL TRIAL: NCT01253096
Title: A Phase II Study of Intratumoral Application of L19IL2 in Patients With Stage III/IV Melanoma.
Brief Title: Intratumoral Application of L19IL2 in Patients With Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2-03/09
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Malignant Melanoma
Keywords: Interleukin; IL2; monoclonal; antibody; cytokine; metastatic; melanoma; tumor targeting; intratumoral; Malignant melanoma with presence of injectable soft-tissue metastases either in clinical stage III or stage IV without visceral metastases.
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L19IL2 (Experimental)
  Interventions: Drug: Intratumoral injections of L19IL2

INTERVENTIONS:
Drug: Intratumoral injections of L19IL2 — Patients will be treated with intratumoral injections of L19IL2 1-3 x weekly. The maximum cumulative dose per week is 20 MioIU. Treatment duration is up to 20 weeks.

SUMMARY:
Phase II, non-randomized, multicenter, prospective study designed to test the efficacy and safety of intratumorally administered L19IL2 in patients suffering from metastatic melanoma.

DETAILED DESCRIPTION:
Phase II, non-randomized, multicenter, prospective study designed to test the efficacy and safety of intratumorally administered L19IL2. L19IL2 binds with high affinity to the EDB domain of Fibronectin, a marker of angiogenesis which is strongly upregulated in malignant melanoma lesions. This binding leads to an increased residence time of the protein at the site of disease. The biologic effect of the IL2 moiety is identical to the one of free IL-2.

The study treatment is up to 20 MioIU L19IL2 per week in patients suffering from histopathologically-proven malignant melanoma with presence of injectable soft-tissue metastases either in clinical stage III or stage IV M1a without visceral metastases. The duration of treatment could be up to 20 weeks. After the end of study visit follow-up is performed every 6 weeks until 12 months from enrollment of each patient.

Tumor assessment will be performed within 2 weeks before start of treatment and at week 12 using immune-related response criteria and RECIST 1.1. To assure that patients do not develop visceral metastases under treatment, an additional tumor assessment will be performed already at week 6 after start of therapy. Assessments at week 24 and 36 will be performed according to RECIST vs. 1.1 criteria only.

Treatment emergent adverse events will be summarized by Common Toxicity Criteria (version 4.02, CTCAE) and worst grade for all treated patients. Laboratory values and change in vital signs will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven malignant melanoma.
* Presence of measurable and injectable soft tissue metastases either in clinical stage III or stage IV M1a.
* Males or females, age >/= 18 years.
* Either without, or after one line of prior systemic treatment for metastatic disease.
* ECOG performance status < 2.
* LDH < 2 x the upper limit of normal.
* Life expectancy of at least 12 weeks.
* Absolute neutrophil count > 1.5 x 10^9/L.
* Hemoglobin > 9.0 g/dL.
* Platelets > 100 x 10^9/L.
* Total bilirubin ≤ 30 µmol/L (or ≤ 2.0 mg/dl).
* ALT and AST ≤ 2.5 x the upper limit of normal (ULN) (5.0 x ULN for patients with hepatic involvement with tumor).
* Serum creatinine < 1.5 x ULN.
* All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v4.02) Grade ≤ 1 unless otherwise specified above.
* Negative serum pregnancy test (for women of child-bearing potential only) at screening.
* If of childbearing potential, agreement to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug.
* Able to provide written Informed Consent.
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Primary ocular melanoma.
* Presence of visceral metastases at screening.
* Evidence of active brain metastases at screening.
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (TA, Tis & Ti) or any cancer curatively treated < 5 years prior to study entry.
* History of HIV infection or infectious hepatitis B or C.
* Presence of active infections (e.g. requiring antimicrobial therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
* Inadequately controlled cardiac arrhythmias including atrial fibrillation.
* Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
* Uncontrolled hypertension.
* Ischemic peripheral vascular disease (Grade IIb-IV).
* Severe diabetic retinopathy.
* Active autoimmune disease.
* History of organ allograft or stem cell transplantation.
* Recovery from major trauma including surgery within 4 weeks prior to administration of study treatment.
* Known history of allergy to IL2, or other intravenously administered human proteins/peptides/antibodies.
* Breast feeding female.
* Anti-tumor therapy within 4 weeks of the administration of study treatment (except small surgery).
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment.
* Planned administration of growth factors or immunomodulatory agents within 7 days before the administration of study treatment.
* Patients in need of systemic treatment for rapidly progressive systemic disease during study treatment and up to 2 weeks after injection of L19IL2.
* Patient requires, or is taking, corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
* Any condition, that in the opinion of the investigator could hamper compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Rate of patients with complete response (CR) of L19IL2 treated Index/Non-Index lesions at week 12 . | week 12

SECONDARY OUTCOMES:
Safety of intratumoral administration of L19IL2 | 1-29 days
Rate of patients with complete response (CR), partial response (PR) and stable disease (SD) of L19IL2 treated Index/Non-Index lesions at week 12. | week 12
Duration of objective response and disease control of L19IL2 treated Index/Non-Index lesions | week 6-46
Overall survival (OS) | 1 year
Rate of patients with complete response (CR), partial response (PR) and stable disease (SD)of all metastases | week 12
Objective response rate of all metastases | week 24, week 36
Disease control rate of all metastases | week 24, week 36

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, Prof. M.D., Principal Investigator — University Hospital Tuebingen (Germany)
Locations (3):
- Universitätsklinik Graz, Graz, Austria
- Germany (2):
  - Medizinischen Hochschule Hannover, Hanover
  - University Hospital, Tübingen